CLINICAL TRIAL: NCT01693718
Title: A Multicenter Phase II Study of Intensive Concomitant Chemoradiotherapy With Filgrastim (GCSF) for Patients With Locoregionally Advanced Head and Neck Cancer
Brief Title: A Multicenter Study of Intensive Concomitant Chemoradiotherapy With Filgrastim (GCSF) for Patients With Locoregionally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12141B
Record Dates: First submitted 2010-08-20; First posted 2012-09-26 (Estimated); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck
Keywords: cancer; advanced; oral cavity; larynx
MeSH Terms: conditions — Neoplasms; Laryngeal Diseases | interventions — Hydroxyurea; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea at 1gm(PO)12hrs x 11days(2gm/day). The first daily dose of hydroxyurea on days 1-5 is given 2 hrs prior to the first fraction of daily radiotherapy.
Drug: 5- Fluorouracil — Start continuous infusion of 5-Fluorouracil at 800mg/m2/day x 5 days (120 hrs.
  Radiation therapy is administered twice daily at 150 cGY per fraction, every other week with chemotherapy.
Drug: Cisplatin — Cisplatin 100mg/m2 I.V. on the evening of the day 1, on cycles 1,3,and 5 only in 200cc NS IV over 2 h. Ensure adequate hydration to keep urine output > 100 cc/ hour.

SUMMARY:
The goal of the study is to test a particular combination of drugs and determine their ability to completely eliminate head and neck cancer.

ELIGIBILITY:
Eligibility Criteria:

1. Patients with Stage IV carcinoma of the nasal or oral cavity, nasopharynx pharynx, larynx, paranasal sinuses, cervical esophagus, or hypopharynx are eligible. Patients with Stage III carcinoma of the nasopharynx, base of tongue and hypopharynx are also eligible. Therapy is given with curative intent.

   Prior to entry in the study the resectability and standard treatment options for each patient will be determined during a joint evaluation by a team composed of an attending surgeon, a radiation oncologist and a medical oncologist. In addition the timing and feasibility of surgery will be determined in each patient prior to initiation of therapy. The unequivocal demonstration of distant metastasis confers in eligibility.
2. Measurable disease is not required, but all disease will be carefully evaluated.
3. Patients must have a histologically or cytologically confirmed diagnosis of squamous cell carcinoma or lymphoepithelioma.
4. Patients must have not received prior chemotherapy or radiotherapy.
5. Patients must have performance status of >60%
6. Patients must have a WBC count of >3.5, an ANC count >1500 and a platlet count of >100,000.
7. The serum creatinine must be equal to or less than 1.5 m/dlor the calculated creatinine clearance must exceed 50cc/min.
8. Patient must be free of significant infection or other severe complicating medical illness.
9. Pregnancy will constitute an absolute contraindication to entrance on this protocol. Females of child-bearing age should be using adequate contraception.

Min Age: 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-03; Primary Completion 2003-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Response Rates | 2-5 years
  To evaluate the activity of 5 cycles of C-FHX/G-CSF in previously untreated patients with stage II and IV locoregionally advanced head and neck cancer.

SECONDARY OUTCOMES:
Feasibility of administering adjuvant CRA and interferon alfa2a | 2-5 years
  To determine the feasibility of administering adjuvant CRA and interferon alfa2a for up to one or until tumor progression in patients completing local therapy.
Side effects of study regimen | 2-5 years
  To determine the pattern and degree of clinical toxicity of this regimen

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, MD, Principal Investigator — The University of Chicago Medical Center
Locations (1):
- The University of Chicago, Chicago, Illinois, United States